CLINICAL TRIAL: NCT06542809
Title: Evaluation of the Propensity of Patients Under rhGH to Envision a Modification of Their Treatment Regimen Toward LAGH
Acronym: TOWARD-LAGH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: The Belux Society for Pediatric Endocrinology and Diabetology (BELSPEED) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024/21FEV/083
Record Dates: First submitted 2024-07-25; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Growth Hormone Deficiency
Keywords: Growth Hormone; New treatment; Propensity; Pediatric
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Belgian and Luxembourgish patients currently under rhGh treatment (Experimental): Patient population studied are Belgian and Luxembourgish patients currently under rhGh treatment in its various official indications (as per the Belgian RIZIV/INAMI monitor : growth hormone deficiency, Turner Syndrome, chronic renal insufficiency, Prader-Willi syndrome, Small for gestational age, Noonan Syndrome, SHOX gene deficiency) and included in the BELGROW Registry Number.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Recruitment will take place through routine paediatric endocrinology consultations with physicians registered with BELSPEED. These doctors will take the time to explain the questionnaire. And allow the patient to complete it.

SUMMARY:
Daily subcutaneous injections of rhGH can be burdensome for patients, leading to poor adherence and reduced growth outcomes. This has spurred the development of long-acting GH (LAGH) analogues that allow for weekly, biweekly, or monthly injections. Previous studies on LAGH analogues have demonstrated their non-inferiority compared to daily rhGH in terms of increasing growth velocity and improving body composition in children and adults with growth hormone deficiency (GHD), respectively, without significant and unexpected adverse events. Since 2020, three molecules have received approval from the Food and Drug Administration (FDA) for the treatment of pediatric GHD: lonapegsomatropin, somatrogon, and somapacitan. These LAGH analogues may offer better patient acceptance, improved tolerance, and greater therapeutic flexibility. However, these LAGH analogues could also be associated with potential clinical issues in terms of therapeutic monitoring, incidence and duration of side effects, and long-term safety due to a non-physiological GH profile. The introduction of these new LAGH products will require clinicians to identify optimal candidates for LAGH therapy and gain knowledge on monitoring and adjusting treatment.

ELIGIBILITY:
Inclusion Criteria:

* Belgian and Luxembourgish patients currently under rhGh treatment in its various official indications (as per the Belgian RIZIV/INAMI monitor : growth hormone deficiency, Turner Syndrome, chronic renal insufficiency, Prader-Willi syndrome, Small for gestational age, Noonan Syndrome, SHOX gene deficiency) and included in the BELGROW Registry
* Male -female
* 0-18 years
* Free written or e-consent and oral consent

Exclusion Criteria:

* No exclusion criteria

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate families and patients propensity with a questionnaire to envision a switch from rhGH treatment to LAGH | Baseline
  By distributing a questionnaire designed by the investigators, they are looking to know if patients and families are already aware of these new treatments, likelihood to improve adherence with LAGH or other benefits they might expect from it, potential to increase/decrease risk of treatment-related side effects, concerns they might have in changing the current treatment, what information would they want to receive from their practitioner.

SECONDARY OUTCOMES:
Evaluate if families/patients response varies according to age, indication of rhGH treatment, any underlying pathology, and/or duration of rhGH treatment. | Baseline
  By distributing a questionnaire designed by the investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lysy, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Woluwe-saint-lambert, Belgium

IPD SHARING:
Plan to Share IPD: No